CLINICAL TRIAL: NCT06970171
Title: Acceptance and Side Effects of Two Different Mandibular Advancement Devices (MADs) in the Treatment of Obstructive Sleep Apnea Syndrome (OSAS)
Brief Title: Acceptance of Mandibular Advancement Devices
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Principal Investigator, Olaf Bernhardt, Prof. Dr. med. dent., University Medicine Greifswald
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MAD08042025
Record Dates: First submitted 2025-04-22; First posted 2025-05-14 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: Obstructive Sleep Apnea Syndrome (OSAS)
Keywords: acceptance; side effects; mandibular advancement device; clinical intervention; treatment
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients randomly selected for arm 1 MAD treatment (Experimental): Patients with primary snoring or with a medical indication for MAD therapy due to OSAS. Patients age must be ≥ 18 and ≤ 75 years. Patients must have a mandibular advancement of at least 5 mm possible (titration starts at 5 mm). Patients must have at least 8 teeth or 4 implants per jaw or with fixed prosthetics or stable removable partial dentures, bilateral support extending to at least the second premolars.
  Interventions: Device: MAD of the Scheu Dental type with lateral guidance wings (MAD-1)
- Patients randomly assigned to arm 2 MAD treatment. (Active Comparator): Patients with primary snoring or with a medical indication for MAD therapy due to OSAS. Patients age must be ≥ 18 and ≤ 75 years. Patients must have a mandibular advancement of at least 5 mm possible (titration starts at 5 mm). Patients must have at least 8 teeth or 4 implants per jaw or with fixed prosthetics or stable removable partial dentures, bilateral support extending to at least the second premolars.
  Interventions: Device: MAD of the Panthera X3 type with lateral guidance wings (MAD-2)

INTERVENTIONS:
Device: MAD of the Scheu Dental type with lateral guidance wings (MAD-1) — The vertical dimension is raised to achieve an incisal edge distance (IED) of 5 mm using a George Gauge, with a mandibular advancement of 5 mm at insertion, progressing to final titrated advancement during the treatment phase.
  Arms: Patients randomly selected for arm 1 MAD treatment
Device: MAD of the Panthera X3 type with lateral guidance wings (MAD-2) — The vertical dimension is raised to achieve a minimum 2 mm interocclusal cusp distance and the lowest possible IED, with a mandibular advancement of 5 mm at insertion, progressing to final titrated advancement during the treatment phase.
  Arms: Patients randomly assigned to arm 2 MAD treatment.

SUMMARY:
Background: Obstructive sleep apnea syndrome (OSAS) is a prevalent condition with significant comorbidities. Mandibular advancement devices (MADs) are an established alternative for patients intolerant to continuous positive airway pressure (CPAP) therapy. However, potential side effects, particularly within the craniomandibular system, warrant further investigation.

Objective: This randomized controlled Phase IV trial aims to compare two different MAD designs (UPS-1 by Scheu Dental and UPS-2 by Panthera X3) in terms of patient acceptance, wearing comfort, adherence, and side effects, especially occlusal changes and temporomandibular discomfort, in OSAS patients over a 12-month period.

Methods: Twenty-eight patients will be stratified by sex and randomized 1:1 into two treatment groups. Assessments include acceptance of the MAD, clinical and digital occlusal analysis (GEDAS), functional examination (DC/TMD), sleep parameters (AHI, ESS, DI), and patient-reported outcomes. Follow-ups were scheduled at 4 weeks, 6 months, and 12 months post-insertion. Data were collected using standardized CRFs and validated questionnaires. Statistical analysis was based on ordinal regression and intention-to-treat and per-protocol populations.

Results & Conclusion: This study will provide evidence on the comparative efficacy and tolerability of two distinct MAD systems, contributing to improved treatment selection in personalized OSAS management.

DETAILED DESCRIPTION:
Partial obstruction of the upper airway during sleep leads to snoring in approximately 40% of men and 24% of women. Epidemiological studies indicate that 50% of these individuals suffer from obstructive sleep apnea syndrome (OSAS) (1, 2).

Sleep-related breathing disorders (SRBD), particularly OSAS, are among the most common causes of non-restorative sleep and sleep disorders. Characteristic patterns include apneas and hypopneas, which may occur with or without pharyngeal obstruction and hypoventilation. Depending on the type of breathing disorder, they may be associated with hypoxemia and can lead to hypercapnia or acidosis.

The consequences of obstructive pharyngeal narrowing are far-reaching. Studies have demonstrated that patients with OSAS frequently experience comorbidities such as neurological disorders, myocardial infarctions, dementia, cardiovascular diseases, and higher mortality rates (3-8). Sleep fragmentation due to nocturnal breathing disturbances and arousals may result in daytime sleepiness and impaired concentration. In the long term, untreated apneas and arousals increase the risk of arterial hypertension, stroke, myocardial infarction, diabetes mellitus, and reduced libido.

Therapeutic options during sleep include continuous positive airway pressure (CPAP) therapy, mandibular advancement devices (MADs), positional therapy, weight reduction, surgical interventions in the ENT region, bimaxillary or mandibular osteotomies, and hypoglossal nerve stimulation.

The choice of therapy depends on the severity of OSAS. For mild to moderate OSAS, MADs, positional therapy, and weight loss are viable options. In severe OSAS, CPAP therapy remains the gold standard. Osteotomies, offering effects comparable to CPAP, and hypoglossal nerve stimulation are reserved for specific clinical cases. In certain cases, a multimodal approach, including surgical methods, may be appropriate regardless of OSAS severity.

CPAP therapy can be delivered as continuous positive airway pressure (CPAP) or automatic positive airway pressure (APAP) (9). However, up to 50% of patients are non-adherent to long-term PAP therapy. For these patients, MADs present a feasible alternative (10). Although MADs are less effective than PAP therapy in reducing the apnea-hypopnea index (AHI) across all OSAS severities, they are similarly effective in mild to moderate cases and are generally preferred by patients (10, 11).

Given the diversity of treatment options, interdisciplinary collaboration among sleep specialists, ENT physicians, and specialized dentists is essential. All treatment measures should be monitored via ambulatory polygraphy or inpatient/semistationary polysomnography.

Prolonged mandibular advancement during sleep may cause symptoms similar to those observed in temporomandibular disorders (TMD), including pain or tension in the masticatory and cranial muscles or in the temporomandibular joints. Asymptomatic events may lead to reversible or irreversible muscle contractures, resulting in occlusal changes, such as bilateral posterior open bite (POB). A study by Perez et al. reported an increase in POB within two years of MAD use (n = 85) (12). The SHIP study found that a POB of more than 3 mm is often associated with TMD symptoms (13). Changes in anterior tooth angulation were observed in patients using MADs (14). Further studies have shown proclination of the upper incisors and labial tipping of lower incisors during MAD therapy (15, 16).

This study aims to assess acceptance, adherence, and potential side effects within the cranio-mandibular system associated with nightly MAD use over a one-year period. Two appliances differing in construction, material and vertical dimension are compared: MAD-1 with lateral wings by Scheu Dental, and MAD-2 with lateral wings by Panthera.

Research Question / Working Hypothesis The objective of this study is to compare two established medical device therapies in a randomized and controlled trial in patients with primary snoring and OSAS with regard to acceptance of the prescribed MAD and adverse effects in terms of splint-related dysfunctions of the cranio-mandibular system and occlusal changes.

Working hypotheses:

1. MAD-1 results in significantly lower patient acceptance compared to MAD-2 (primary endpoint).
2. MAD-1 leads to a significantly higher number of pressure-sensitive areas in the masticatory muscles and temporomandibular joints than MAD-2.
3. MAD-1 is associated with significantly more head pain than MAD-2.
4. A higher loss of posterior contact points is observed in MAD-1 than in MAD-2.
5. The extent of protrusion and vertical dimension after titration and after 12 months is lower in MAD-2 compared to MAD-1.
6. MAD-1 and MAD-2 do not differ significantly in terms of sleep parameters: ESS, AHI, desaturation index (DI), and mean oxygen saturation.

Recruitment Description: Patients are recruited at the Center for Dentistry, Oral and Maxillofacial Medicine and examined by staff specialized in treating OSAS patients using MADs, in collaboration with referring sleep medicine centers.

Investigator Calibration All study dentists will be trained and calibrated by the study director in the examination tools and data collection before study initiation. The training center is the Department of Restorative Dentistry, Periodontology, and Endodontology. On April 8, 2025, both study dentists were briefed on the examination procedure and the administration of the questionnaires. In addition, clinical functional analysis will be demonstrated.

Sleep Medicine Examination Patients were referred to the Center for Dentistry, Oral and Maxillofacial Medicine at the University Medical Center Greifswald for fabrication and insertion of a MAD, based on prior diagnosis by a sleep medicine specialist for the treatment of OSAS or snoring.

Baseline Examination Anamnesis will be performed, followed by assessment of dental status and the Periodontal Screening Index (PSI) to verify eligibility for MAD therapy. A functional status evaluation, clinical and digital occlusion protocols (GEDAS), the Graded Chronic Pain Scale (GCPS) and Epworth Sleepiness Scale (ESS) will be recorded.

Functional status is assessed using the standardized DC/TMD protocol. All questionnaires are based on validated recommendations. The examination procedures are part of routine diagnostics, standardized across participating dental practices for this study.

Block randomization (1:1 ratio) is conducted in a decentralized manner using sealed envelopes, each containing the allocation key for the respective MAD. The allocation is stratified by sex, as sex is a strong predictor for both sleep disorders and temporomandibular dysfunctions.

The upper and lower jaws are scanned to fabricate the respective therapeutic devices, and protrusive bite registrations are taken (Trios, 3Shape Germany GmbH). The starting position for mandibular advancement is standardized at 5 mm. These scans are provided to patients free of charge as a benefit for study participation.

Insertion of MAD (Start of Therapy) and Follow-up After One Week The lab-fabricated splint (MAD-1 or MAD-2) is inserted (with an initial mandibular advancement of 5 mm) and checked for proper fit. Particular attention is given to uniform contact between the upper and lower components and a tension-free seat on the dentition. Interferences are selectively adjusted if necessary. Patients are instructed to wear the device consistently during sleep.

All patients receive detailed instructions for jaw exercises to be performed each morning after waking and in the evening before going to sleep.

First Follow-up Visit (4 Weeks After Insertion) Four weeks after insertion, the titration phase begins. This involves the gradual adjustment of mandibular advancement to optimize sleep-related parameters while minimizing unwanted side effects. The advancement is increased until optimal clinical and sleep-related outcomes are reached, or until further advancement becomes intolerable for the patient.

The functional status, occlusion protocol, ESS questionnaire and an assessment of wearing comfort are reassessed.

Second Follow-up Visit (6 Months After Start of Therapy) Six months after therapy initiation, another follow-up appointment is conducted to reassess the functional status, occlusion protocol, the ESS questionnaire, an assessment of wearing comfort.

Third Follow-up Visit (12 Months After Start of Therapy) The third follow-up takes place 12 months after the start of therapy. The functional status, ESS questionnaire, occlusion protocol, assessment of wearing comfort and bite registration for scanning and contact point analysis (GEDAS, Greifswald Digital Analyzing System) are collected.

A patient may only be enrolled in the study after providing informed consent, having been adequately informed-both verbally and in writing-by a study dentist about the nature, scope, and implications of the study.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication for MAD therapy due to OSAS
* Mandibular advancement of at least 5 mm possible
* Fixed prosthetics or stable removable partial dentures
* Bilateral support extending to at least the second premolars
* Legal capacity and signed informed consent

Exclusion Criteria:

* Polyarthritis
* Mouth opening < 30 mm
* More than two prior therapy attempts
* Fibromyalgia, neuralgia
* Central sleep apnea syndrome
* Pulmonary diseases
* Untreated generalized periodontitis
* Chronic dysfunctional pain (GCPS Grade 3-4)
* Long-term use of psychotropic or analgesic medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-05-05 (Estimated); Primary Completion 2027-05-05 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the MAD | 4 weeks, 6 months, 12 months
  wearing comfort of the MAD, assessed using a numeric rating scale (NRS; 0-10) at follow-up time points

SECONDARY OUTCOMES:
Orofacial Pain | 4 weeks, 6 months, 12 months
  Change of pain in the orofacial region measured by numeric rating scale (NRS, 0-10)
Pressure Pain in the Temporomandibular Joint and Masticatory Muscles | 4 weeks, 6 months, 12 months
  Change in number of pressure-sensitive points during palpation of masticatory muscles and TMJs
Number of Posterior Contact Points | 4 weeks, 6 months, 12 months
  change of the number of occluding posterior teeth
GEDAS (Greifswald Digital Analyzing System) | 12 months
  Digital occlusion protocol assessed via occlusal records in habitual intercuspation; evaluated using GEDAS (Greifswald Digital Analyzing System) based on transparent contact areas

OTHER OUTCOMES:
Epworth Sleepiness Scale (ESS) | 4 weeks, 6 months, 12 months
  Change in daytime sleepiness measured by Epworth Sleepiness Scale. ESS is a short questionnaire for the detection of daytime sleepiness. (ESS, 0-24, <11 no daytime sleepiness)
Apnea-Hypopnea Index (AHI) | 12 months
  The Apnea-Hypopnea Index (AHI) is a metric indicating the number of apneas and hypopneas a patient experiences during sleep. It is determined through polysomnographic recording in a sleep laboratory. Based on the AHI value, sleep apnea is classified as mild, moderate, or severe.
Desaturation Index (DI) | 12 months
  The Desaturation Index (DI) refers to the number of oxygen desaturation events per hour of sleep.
Mean Oxygen Saturation | 12 months
  Mean oxygen saturation during sleep

CONTACTS AND LOCATIONS:
Overall Officials: Olaf Bernhardt, Prof. Dr. med.dent., Principal Investigator — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Department of Restorative Dentistry, Periodontology and Endodontology, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abe S, Huynh NT, Romprss PH, de Grandmont P, Landry-Schonbeck A, Landry ML, Kato T, Kawano F, Lavigne GJ. Sleep Quality and Comfort Reported by Sleep Bruxism Individuals Wearing the Occlusal Splint and Mandibular Advancement Splint: Revisiting Two Crossover Studies. Int J Prosthodont. 2023 May;36(2):138-147. doi: 10.11607/ijp.7525. Epub 2023 May 24. PMID 36484654
- [Background] Uniken Venema JAM, Doff MHJ, Joffe-Sokolova DS, Wijkstra PJ, van der Hoeven JH, Stegenga B, Hoekema A. Dental side effects of long-term obstructive sleep apnea therapy: a 10-year follow-up study. Clin Oral Investig. 2020 Sep;24(9):3069-3076. doi: 10.1007/s00784-019-03175-6. Epub 2019 Dec 20. PMID 31863188
- [Background] Doff MH, Hoekema A, Pruim GJ, Huddleston Slater JJ, Stegenga B. Long-term oral-appliance therapy in obstructive sleep apnea: a cephalometric study of craniofacial changes. J Dent. 2010 Dec;38(12):1010-8. doi: 10.1016/j.jdent.2010.08.018. Epub 2010 Sep 8. PMID 20831889
- [Background] Fransson AM, Svenson BA, Isacsson G. The effect of posture and a mandibular protruding device on pharyngeal dimensions: a cephalometric study. Sleep Breath. 2002 Jun;6(2):55-68. doi: 10.1007/s11325-002-0055-7. PMID 12075480
- [Background] Gesch D, Bernhardt O, Kocher T, John U, Hensel E, Alte D. Association of malocclusion and functional occlusion with signs of temporomandibular disorders in adults: results of the population-based study of health in Pomerania. Angle Orthod. 2004 Aug;74(4):512-20. doi: 10.1043/0003-3219(2004)0742.0.CO;2. PMID 15387030
- [Background] Perez CV, de Leeuw R, Okeson JP, Carlson CR, Li HF, Bush HM, Falace DA. The incidence and prevalence of temporomandibular disorders and posterior open bite in patients receiving mandibular advancement device therapy for obstructive sleep apnea. Sleep Breath. 2013 Mar;17(1):323-32. doi: 10.1007/s11325-012-0695-1. Epub 2012 Apr 4. PMID 22477031
- [Background] Gislason T, Janson C, Vermeire P, Plaschke P, Bjornsson E, Gislason D, Boman G. Respiratory symptoms and nocturnal gastroesophageal reflux: a population-based study of young adults in three European countries. Chest. 2002 Jan;121(1):158-63. doi: 10.1378/chest.121.1.158. PMID 11796445
- [Background] Pelttari L, Rauhala E, Polo O, Hyyppa MT, Kronholm E, Viikari J, Kantola I. Upper airway obstruction in hypothyroidism. J Intern Med. 1994 Aug;236(2):177-81. doi: 10.1111/j.1365-2796.1994.tb01280.x. PMID 8046317
- [Background] Tingting X, Danming Y, Xin C. Non-surgical treatment of obstructive sleep apnea syndrome. Eur Arch Otorhinolaryngol. 2018 Feb;275(2):335-346. doi: 10.1007/s00405-017-4818-y. Epub 2017 Nov 24. PMID 29177626
- [Background] Mohsenin V. Is sleep apnea a risk factor for stroke? A critical analysis. Minerva Med. 2004 Aug;95(4):291-305. PMID 15334043
- [Background] Gottlieb DJ, Chase C, Vezina RM, Heeren TC, Corwin MJ, Auerbach SH, Weese-Mayer DE, Lesko SM. Sleep-disordered breathing symptoms are associated with poorer cognitive function in 5-year-old children. J Pediatr. 2004 Oct;145(4):458-64. doi: 10.1016/j.jpeds.2004.05.039. PMID 15480367
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Lugaresi E, Cirignotta F, Coccagna G, Piana C. Some epidemiological data on snoring and cardiocirculatory disturbances. Sleep. 1980;3(3-4):221-4. doi: 10.1093/sleep/3.3-4.221. No abstract available. PMID 7221330
- [Background] Cook RJ, Farewell VT. On multiplicity considerations in the design and analysis of clinical trials. J Roy Statist Soc 1996;159:93-110.
- [Background] Ringqvist M, Walker-Engstrom ML, Tegelberg A, Ringqvist I. Dental and skeletal changes after 4 years of obstructive sleep apnea treatment with a mandibular advancement device: a prospective, randomized study. Am J Orthod Dentofacial Orthop. 2003 Jul;124(1):53-60. doi: 10.1016/s0889-5406(03)00240-3. PMID 12867898
- [Background] Haviv Y, Rettman A, Aframian D, Sharav Y, Benoliel R. Myofascial pain: an open study on the pharmacotherapeutic response to stepped treatment with tricyclic antidepressants and gabapentin. J Oral Facial Pain Headache. 2015 Spring;29(2):144-51. doi: 10.11607/ofph.1408. PMID 25905532
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728